CLINICAL TRIAL: NCT06255106
Title: Comparative Computed Tomography Analysis of the Cast Index and Three-Point Index in Distal Radius Fracture Treatment
Brief Title: CT Analysis Comparing Cast and Three-Point Indexes in Distal Radius Fracture Care
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yasar Samet Gokceoglu, Principal investigator, Istanbul University
Other Study IDs: DistalRadiuscast
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Distal Radius Fractures
Keywords: distal radius fracture; cast index; three point index; computed tomography
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Group 1, consisting of individuals treated with a cast
  Interventions: Other: cast treatment
- Group 2: Group 2, comprising those who underwent surgical intervention (Open reduction volar plate fixation.
  Interventions: Other: cast treatment

INTERVENTIONS:
Other: cast treatment — Surgical intervention vs cast treatment
  Other Names: Open reduction volar plate fixation

SUMMARY:
Objectives: To compare the cast index and three-point index measurements obtained using computed tomography (CT) with those acquired using conventional methods for treating distal radius fractures Design: A retrospective cohort study Setting: Level 1 trauma center Patients: One hundred and thirteen (45 men and 68 women) patients with distal radius fractures Interventions: Patients with distal radius fractures were retrospectively analyzed and received either conservative cast treatment or surgical intervention through open reduction and internal fixation between 2016 and 2022.

Main outcome measurements: The study evaluated the cast index and three-point index in the cast-treated group and their effectiveness using the Sarmiento index. Furthermore, radial height, volar tilt, and radial inclination were compared between the surgically treated and cast-treated groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Diagnosed with distal radius fracture
* Treated with either cast or volar plate osteosynthesis were included in the study.

Exclusion Criteria:

* Patients with multiple fractures in the same upper extremity
* Those treated with dorsal plates or external fixators
* Individuals with open fractures
* Patients with known systemic or rheumatologic diseases
* Those with cervical disk problems
* Individuals lacking post-cast removal CT data
* Patients with incomplete medical records were excluded.

Ages: 19 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with distal radius fractures.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Radial height | 2 weeks
  Radiologic outcome measurement
Radial İnclination | 2 weeks
  Radiologic outcome measurement
Volar tilt | 2 weeks
  Radiologic outcome measurement
Sarmiento radiological score | 2 weeks
  success of cast treatment

SECONDARY OUTCOMES:
Axial Cast İndex | 2 weeks
  Cast index measure in axial plane CT
Three point index CT | 2 weeks
  Three point index measure in CT

CONTACTS AND LOCATIONS:
Overall Officials: Yaşar Samet Gökçeoğlu, MD, Principal Investigator — Istanbul University
Locations (1):
- University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song J, Yu AX, Li ZH. Comparison of conservative and operative treatment for distal radius fracture: a meta-analysis of randomized controlled trials. Int J Clin Exp Med. 2015 Oct 15;8(10):17023-35. eCollection 2015. PMID 26770293
- [Background] Kahraman HC, Sibar K, Alemdaroglu KB, Subasi IO, Gokgoz MB. Is three-point index reliable in the follow-up of the distal radius metaphys fractures in the pediatric age group? J Pediatr Orthop B. 2023 Jul 1;32(4):369-377. doi: 10.1097/BPB.0000000000001032. Epub 2022 Nov 14. PMID 36377954
- [Result] Owen RA, Melton LJ 3rd, Johnson KA, Ilstrup DM, Riggs BL. Incidence of Colles' fracture in a North American community. Am J Public Health. 1982 Jun;72(6):605-7. doi: 10.2105/ajph.72.6.605. PMID 7072880
- [Result] Alemdaroglu KB, Iltar S, Aydogan NH, Say F, Kilinc CY, Tiftikci U. Three-point index in predicting redisplacement of extra-articular distal radial fractures in adults. Injury. 2010 Feb;41(2):197-203. doi: 10.1016/j.injury.2009.08.021. Epub 2009 Sep 26. PMID 19782974
- [Result] Hosseinzadeh P, Olson D, Eads R, Jaglowicz A, Goldfarb CA, Riley SA. Radiologic Evaluation of the Distal Radius Indices in Early And Late Childhood. Iowa Orthop J. 2018;38:137-140. PMID 30104936